CLINICAL TRIAL: NCT02313480
Title: Does the Addition of Massage to Manual Therapy and Exercise Improve Outcome in Chronic Neck Pain?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Society of Musculoskeletal Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RM01
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- non-massage group (Active Comparator): received exercise, manual therapy and advice over the 30 minute intervention period, in conjunction with an exercise program to perform at home.
  Interventions: Other: massage
- massage group (Experimental): Received massage, exercise, manual therapy and advice over the 30 minute intervention period, in conjunction with an exercise program to perform at home.
  Interventions: Other: massage

INTERVENTIONS:
Other: massage — Swedish massage was included in one arm of the study and not the other. Administered by a trained therapist as part of the usual 30 minute treatment time. Amount of massage administered dependant on Therapist's clinical reasoning

SUMMARY:
To date, the benefits of massage in chronic neck pain patients has only been investigated as a singular treatment, rather than as part of a treatment package. The need for this research has been highlighted in the literature (Ezzo et al, 2007; Haraldsson et al, 2006) This research aimed to establish whether the addition of massage to a program of exercise and manual therapy offers any additional benefits over exercise and manual therapy alone in the treatment of patients with chronic neck pain.

DETAILED DESCRIPTION:
39 patients with neck pain of greater than three months duration were randomised to either a massage or non-massage group in a primary care setting in the Dublin region. One therapist administered all treatments. Randomisation was carried out by the use of sequential sampling, utilising permuted blocks. Patients were excluded from the study if they had severe co-existing disease, had neck pain due to fracture, tumour, infection or other non-mechanical causes, or if the patient had a diagnosis of osteoporosis anywhere in the body.

Both groups underwent up to eight weekly physiotherapy sessions. The non-massage group received exercise, manual therapy and advice over the 30 minute intervention period, in conjunction with an exercise program to perform at home. The massage group received all of the above as well as Swedish massage. Follow up was for the duration of treatment only.

A number of T-tests and non-parametric tests were conducted to establish if the two groups were comparable at baseline.

A mixed ANOVA was then used to analyse between-group and within-group data simultaneously. No blinding was possible, although the questionnaires were self-administered which may have limited bias.

ELIGIBILITY:
Inclusion Criteria:

* neck pain for greater than three months
* over 18 years of age
* had not received treatment for their neck pain in the previous month
* could speak conversational English
* were not involved in any current compensation case and
* had provided written, informed consent.

Exclusion Criteria:

* severe co-existing disease,
* neck pain due to fracture, tumour, infection or other non-mechanical causes,
* if the patient had a diagnosis of osteoporosis anywhere in the body.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale | Compared baseline to score after 8 weeks of treatment
  Used to accurately measure pain. On this, patients verbally rated their usual and worst (in the last week) pain from 0 ("no pain") to 10 ("worst possible pain"). Its test-retest reliability in the chronic neck pain population was established as fair to moderate (intraclass correlation coefficient (ICC) =.76; 95% CI, .51-.87) by Cleland et al (2008). Farrar et al (2010) found a difference of two points to be a clinically meaningful change in the chronic pain population.

SECONDARY OUTCOMES:
Neck Disability Index | Compared baseline to score after 8 weeks of treatment
  The NDI (Appendix 3) is the most widely used and most strongly validated instrument for assessing self-rated disability in patients with neck pain (Vernon, 2008).It includes ten self-report items covering activities of daily living, concentration and pain. Responses are on a 0-5 point scale, with a total score ranging from 0 (no pain or disability) to 50 (severe pain and disability; Gay et al, 2007).

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Atkins, Physio, Study Chair — Society of Musculoskeletal Medicine

REFERENCES:
- [Background] Ezzo J, Haraldsson BG, Gross AR, Myers CD, Morien A, Goldsmith CH, Bronfort G, Peloso PM; Cervical Overview Group. Massage for mechanical neck disorders: a systematic review. Spine (Phila Pa 1976). 2007 Feb 1;32(3):353-62. doi: 10.1097/01.brs.0000254099.07294.21. PMID 17268268
- [Background] Haraldsson BG, Gross AR, Myers CD, Ezzo JM, Morien A, Goldsmith C, Peloso PM, Bronfort G; Cervical Overview Group. Massage for mechanical neck disorders. Cochrane Database Syst Rev. 2006 Jul 19;(3):CD004871. doi: 10.1002/14651858.CD004871.pub3. PMID 16856066
- [Background] Cleland JA, Childs JD, Whitman JM. Psychometric properties of the Neck Disability Index and Numeric Pain Rating Scale in patients with mechanical neck pain. Arch Phys Med Rehabil. 2008 Jan;89(1):69-74. doi: 10.1016/j.apmr.2007.08.126. PMID 18164333
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Vernon H. The Neck Disability Index: state-of-the-art, 1991-2008. J Manipulative Physiol Ther. 2008 Sep;31(7):491-502. doi: 10.1016/j.jmpt.2008.08.006. PMID 18803999
- [Background] Gay RE, Madson TJ, Cieslak KR. Comparison of the Neck Disability Index and the Neck Bournemouth Questionnaire in a sample of patients with chronic uncomplicated neck pain. J Manipulative Physiol Ther. 2007 May;30(4):259-62. doi: 10.1016/j.jmpt.2007.03.009. PMID 17509434